CLINICAL TRIAL: NCT03785106
Title: Implementation for Tuberculosis Preventive Therapy Among Latent Tuberculosis Infection in HIV-infected Individuals Using Novel Regimen of Isoniazid/Rifapentine Daily (4 Weeks) Compared to Isoniazid/Rifapentine Weekly (12 Weeks)
Brief Title: Tuberculosis Preventive Therapy Among Latent Tuberculosis Infection in HIV-infected Individuals
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other); Police General Hospital (Other); Pranangklao Hospital (Unknown); Taksin Hospital (Unknown); Bhumibol Adulyadej Hospital (Other); Klang Hospital (Unknown); Chiang Rai Prachanukroh Hospital (Unknown); Sanpatong Hospital (Unknown); Queen Sawang Vadhana Memorial Hospital (Unknown); Buddhachinnaraj Hospital (Unknown); Maharat Nakhon Ratchasima Hospital (Other); HatYai Hospital (Other); Srinagarind Hospital, Khon Kaen University (Other); Sisaket Hospital (Unknown); The Public Health Centre 28 Krung thon buri (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIV-NAT 255
Record Dates: First submitted 2018-12-19; First posted 2018-12-24 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: HIV-infected Participants With Latent TB Infection in High TB Burden Country
Keywords: people living with HIV (PLHIV)
MeSH Terms: interventions — Isoniazid; Pyridoxine; Vitamin B 6

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, randomized, open-label, phase III clinical trial comparing a 4-week daily INH/RPT regimen (1HP) to a 12-weekly INH/RPT (3HP) for the treatment of LTBI in HIV-infected participants without evidence of active TB.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1HP (Experimental): 4-week daily regimen of weight-based RPT and INH, plus pyridoxine (vitamin B6)
  Interventions: Drug: Isoniazid/Rifapentine daily (4 weeks) plus pyridoxine (vitamin B6)
- 3HP (Active Comparator): 12-weekly INH/RPT regimen, plus pyridoxine (vitamin B6)
  Interventions: Drug: Isoniazid/Rifapentine 12-weekly plus pyridoxine (vitamin B6)

INTERVENTIONS:
Drug: Isoniazid/Rifapentine daily (4 weeks) plus pyridoxine (vitamin B6) — Isoniazid/Rifapentine daily (4 weeks) plus pyridoxine (vitamin B6)
  Arms: 1HP
Drug: Isoniazid/Rifapentine 12-weekly plus pyridoxine (vitamin B6) — Isoniazid/Rifapentine 12-weekly plus pyridoxine (vitamin B6)
  Arms: 3HP

SUMMARY:
The investigators want to know if ultra-short, effective treatment for latent tuberculosis (TB) infection (LTBI) could dramatically reduce the global incidence of active TB or not. The investigators hypothesize that short-course (4-week) daily isoniazid/rifapentine (INH/RPT) (1HP) is not inferior to standard -course (12 weeks) INH/RPT weekly regimen (3HP) for the prevention of TB in human immunodeficiency virus (HIV)-infected individuals.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, open-label, phase III clinical trial comparing a 4-week daily INH/RPT regimen (1HP) to a 12-weekly INH/RPT (3HP) for the treatment of LTBI in HIV-infected participants without evidence of active TB. The primary objective will be efficacy of active TB prevention. The study will also assess safety and tolerability of the regimens, adherence to the treatments, and patterns of antibiotic resistance among Mycobacterium tuberculosis (MTB) isolates in participants who fail on these prophylactic regimens.

Under this study, there is one substudy entitled, "Pharmacokinetic study of rifapentine, dolutegravir, and tenofovir alafenamide in HIV-infected individual with latent tubersulosis infection". There will be a subgroup of patients who will participate in this pharmacokinetic study of rifapentine and dolutegravir (DTG) / tenofovir alafenamide (TAF). Randomization is based on cluster of differentiation 4 (CD4) categories : < 200, 200-350, > 500 cells/mm3 and VL <50 or >50 copies/ml.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV-1 infection by standard HIV test or plasma HIV-1 RNA viral load and received ART within 12 months. Participants received ART more than 12 months would be allowed if CD4 cell counts is less than 350 cells/mm3
2. 18 years and older
3. Evidence of latent TB infection, either by TST ≥5 mm or positive interferon gamma release assay (IGRA) or history of close contact with active pulmonary TB* within 3 months prior entry visit or residing in a high TB burden area** NOTE * close contact is referred to person living/sharing in the same room with active pulmonary TB participants for > 4 hours/day

   ** high TB burden areas are defined as areas with an estimated or reported TB prevalence of 100 to 300/100,000, according to the WHO. Thailand is included in high TB burden areas.
4. Laboratory values obtained within 30 days prior to entry

   * Absolute neutrophil count (ANC) >750 cells/mm3
   * Hemoglobin >7.4 g/dL
   * Platelet count >50,000/mm3
   * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) <3x upper limit of normal (ULN)
   * Total bilirubin <2.5 X ULN
5. Chest radiograph or chest computed tomography (CT) scan without evidence of active tuberculosis, unless one has been performed within 90 days prior to entry.
6. Female participants who are participating in sexual activity that could lead to pregnancy must agree to use one reliable non-hormonal form of contraceptive (i.e., condoms, IUD, diaphragm) during RPT treatment and contraception should be remain to 6 weeks post RPT NOTE Female participants who are not of reproductive potential or whose male partner(s) have undergone successful vasectomy with documented azoospermia or have documented azoospermia are eligible without requiring the use of contraceptives. Participant-reported history is acceptable documentation of menopause, hysterectomy, or bilateral oophorectomy or bilateral tubal ligation.
7. All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization) while receiving RPT and for 6 weeks after stopping this drug.
8. Body weight > 40 kg
9. Ability and willingness of participant to provide informed consent

Exclusion Criteria:

1. Treatment for active or latent TB (pulmonary or extrapulmonary) within 2 years prior to study entry or presence of any confirmed or probable active TB at screening.
2. History of Isoniazid (INH) or Rifampicin (RIF)/Rifabutin (RFB) resistant TB at any time prior to study entry or known exposure to INH or RIF/RFB resistant TB (e.g., household member of a person with MDR or XDR TB) at any time prior to study entry.
3. Treatment for >14 consecutive days with a rifamycin or >30 consecutive days with INH at any time during the 2 years prior to enrollment.
4. Current or planned use of protease inhibitor-based ART.
5. Currently on a salvage ART regimen, defined as a regimen started due to confirmed HIV virologic failure on a prior ART regimen or due to known HIV drug resistance.
6. History of liver cirrhosis at any time prior to study entry.
7. Evidence of acute hepatitis, such as abdominal pain, jaundice, dark urine, and/or light stools within 90 days prior to entry.
8. Diagnosis of porphyria at any time prior to study entry.
9. Peripheral neuropathy ≥Grade 2 according to the Division of AIDS (DAIDS) Toxicity Table, within 90 days prior to study entry.
10. Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation.
11. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
12. Acute or serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry.
13. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2038-03 (Estimated); Study Completion 2038-03 (Estimated)

PRIMARY OUTCOMES:
efficacy in preventing active TB (proportion of participants that do not have active TB by the end of the study) | 3 years
  proportion of participants that do not have active TB by the end of the study
safety of the regimens (proportion of participants that do not have any side effects throughout the study period) | 3 years
  proportion of participants that do not have any side effects throughout the study period
tolerability to the regimens (proportion of participants that can complete the treatment course) | 3 years
  proportion of participants that can complete the treatment course
prevalence of drug resistance of MTB | 3 years
  proportion of participants with drug resistance to MTB

SECONDARY OUTCOMES:
severity of the condition | 3 years
  proportion of participants that have side effects of grade more than or equal to 3 signs
presence of symptoms | 3 years
  proportion of participants that have symptoms during the study period
level of CBC | 3 years
  assess the level of CBC
level of ALT | 3 years
  assess the level of ALT
level of AST | 3 years
  assess the level of AST
level of total bilirubin | 3 years
  assess the level of total bilirubin
level of ALK | 3 years
  assess the level of ALK
level of creatinine | 3 years
  assess the level of creatinine
death | 3 years
  time from randomization to death from any cause (TB and non TB events)
when TB culture becomes positive | 3 years
  how much time does it take to have positive TB culture
when TB is confirmed by clinical examination | 3 years
  how much time does it take to have TB diagnosed via clinical examination
adherence to LTBI treatment | 3 years
  proportion of pills missed during treatment period based on self report
consistency of taking LTBI treatment | 3 years
  proportion of pills missed during treatment period based on clinical assessment
treatment discontinuation | 3 years
  proportion of participants with permanent LTBI treatment discontinuation due to all causes
discontinuation of study due to adverse drug reactions | 3 years
  Proportion of participants that have discontinued the study because of adverse drug reactions
CD4 count | 3 years
  CD4 count at baseline
CD4 count to confirmed or probable TB | 3 years
  CD4 count at time from randomization to culture-confirmed or probable TB
time it takes for TB to be confirmed by IGRA | 3 years
  how much time does it take to confirm TB diagnosis via IGRA
TST result at baseline | day 0
  TST result at day 0

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre
Locations (16):
- Thailand (16):
  - Klang Hospital, Bangkok
  - Bhumibol Adulyadej Hospital, Bangkok
  - HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Police General Hospital, Bangkok
  - Taksin Hospital, Bangkok
  - the Public Health Centre 28 Krung thon buri, Bangkok
  - Sanpatong Hospital, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Queen Savang Vadhana Memorial Hospital, Chon Buri
  - Srinagarind Hospital, Khon Kaen
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima
  - Pranangklao Hospital, Nonthaburi
  - Buddhachinnaraj Hospital, Phitsanulok
  - Sisaket Hospital, Si Sa Ket
  - Hatyai Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: No